CLINICAL TRIAL: NCT01332201
Title: A Phase II, Open Label, Parallel Group, Multi-center Study to Compare the Pharmacokinetics of Tacrolimus in Adult Subjects Undergoing Primary Allograft Transplantation Receiving an Advagraf® or Prograf® Based Immunosuppressive Regimen, Including a Long-term Follow-up
Brief Title: Study to Compare the Pharmacokinetics of Tacrolimus in Adult Transplant Recipients Treated With Advagraf® or Prograf®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PMR-EC-1501; 2010-019859-21 (EudraCT Number)
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Heart Transplantation; Lung Transplantation; Pancreas (Including SPK) Transplantation
Keywords: Advagraf; Heart; Lung; Pancreas; Transplant; Immunosuppression; Pharmacokinetics
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Advagraf (Experimental)
  Interventions: Drug: Advagraf
- Prograf (Active Comparator)
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Advagraf — oral
  Other Names: FK506E; MR4; tacrolimus modified release
  Arms: Advagraf
Drug: Prograf — oral
  Other Names: tacrolimus; FK506
  Arms: Prograf

SUMMARY:
Comparison of tacrolimus blood levels in adults who have received a transplant and are taking either Prograf or Advagraf anti-rejection therapy immediately following surgery. This is followed by checking of safety and effectiveness for one year.

ELIGIBILITY:
Inclusion Criteria:

* must receive first oral dose of tacrolimus one day (lung, pancreas or Simultaneous Pancreas Kidney (SPK) recipients) or three days (heart recipients) after transplantation (skin closure)
* negative pregnancy test prior to enrolment (females)
* agree to practice effective birth control during the study
* treated since transplantation with Antithymocyte globulin/ Mycophenolate Mofetil/steroids (ATG/MMF/steroids), gastric motility resumed and renal function adequate (<230 µmol/l (<2.6 ml/dl)) on Day 1

Exclusion Criteria:

* receiving a multi-organ transplant (with the exception of SPK) or previously received an organ transplant (including re-transplantation)
* pulmonary vascular resistance ≥4 Wood units despite medication
* required an emergency ventricular assist device within one week prior to transplantation
* significant renal impairment
* significant liver disease
* malignancies or a history of malignancy within the last 5 years
* significant, uncontrolled concomitant infections and/or severe diarrhoea, vomiting, active upper gastrointestinal disorder that may affect the absorption of tacrolimus, or active peptic ulcer
* requires systemic immunosuppressive medication for any other indication than transplantation
* diagnosis of cystic fibrosis
* pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
determine steady state systemic exposure (AUC 0-24h) | Day 1, Day 3, Day 7 and Day 42

SECONDARY OUTCOMES:
determine Cmax (maximum concentration) | Day 1, Day 3, Day 7 and Day 42
determine tmax (time to attain Cmax) | Day 1, Day 3, Day 7 and Day 42
determine C24 (concentration prior to next morning dose) | Day 1, Day 3, Day 7 and Day 42
describe rejection episodes | up to 58 weeks
describe subject survival | up to 58 weeks
describe graft survival | up to 58 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe Ltd.
Locations (8):
- Vienna, Austria
- Leuven, Belgium
- Paris, France
- Italy (2):
  - Milan
  - Padua
- Taipei, Taiwan
- United Kingdom (2):
  - London
  - Manchester

REFERENCES:
- See also: Link to results on EudraCT — https://www.clinicaltrialsregister.eu/ctr-search/trial/2010-019859-21/results